CLINICAL TRIAL: NCT00283049
Title: Safety and Efficacy of Insulin Glargine Injection [rDNA Origin] Treatment in Place of the TZD or the Sulfonylurea or Metformin in Triple Agent Therapy for T2DM Adult Subjects With Unsatisfactory Control
Brief Title: Insulin Glargine Injection Treatment in Place of Thiazolidinedione (TZD), Sulfonylurea, or Metformin in Triple Agent Therapy for Type 2 Diabetes Mellitus (T2DM) Adult Subjects With Unsatisfactory Control
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to technical issues relating to the Electronic diary data.
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4052
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2010-02-19 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine

ARMS (3):
- Insulins + Sulfonylurea (SU) + Thiazolidinedione (TZD) (Experimental): Arm 1: Insulin glargine administered subcutaneously once daily plus a sulfonylurea and a TZD. Insulin glulisine will be added after Week 12 or later for those subjects needing prandial insulin therapy (HbA1c >6.5%)
  Interventions: Drug: Insulin Glargine; Drug: Insulin Glulisine
- Insulins + Metformin (MET) + Thiazolidinedione (TZD) (Experimental): Arm 2: Insulin glargine administered subcutaneously once daily plus metformin and a TZD. Insulin glulisine will be added after Week 12 or later for those subjects needing prandial insulin therapy (HbA1c >6.5%)
  Interventions: Drug: Insulin Glargine; Drug: Insulin Glulisine
- Insulins + Metformin (MET) + Sulfonylurea (SU) (Experimental): Arm 3: Insulin glargine administered subcutaneously once daily plus metformin and a sulfonylurea. Insulin glulisine will be added arms after Week 12 or later for those subjects needing prandial insulin therapy (HbA1c >6.5%)
  Interventions: Drug: Insulin Glargine; Drug: Insulin Glulisine

INTERVENTIONS:
Drug: Insulin Glargine — Insulin glargine administered subcutaneously once daily.
Drug: Insulin Glulisine — Insulin glulisine will be added after Week 12 or later for those subjects needing prandial insulin therapy (HbA1c >6.5%)

SUMMARY:
The purpose of this study is to compare the change in hemoglobin A1c (HbA1c) from baseline to Week 12 between the 3 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for enrollment into the study:

1. 18 to 79 years of age, inclusive
2. Diagnosis of type 2 diabetes mellitus
3. Continuous treatment with therapeutic dosages of a thiazolidinedione (rosiglitazone or pioglitazone), metformin, and a sulfonylurea daily prior to entering the study
4. Screening HbA1c ≥ 7.0%
5. Fasting C-peptide concentration ≥ 0.27 ng/ml
6. Negative glutamic acid decarboxylase (GAD) antibodies
7. Demonstrated ability and willingness to perform self-monitoring blood glucose (SMBG) using a plasma-referenced glucose meter and to maintain an electronic diary
8. Demonstrated ability and willingness to use an electronic diary to record SMBG results, insulin doses, and hypoglycemic events.
9. Signed, informed consent and Health Insurance Portability and Accountability Act (HIPAA) documentation

Exclusion Criteria:

1. Stroke, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, or angina pectoris, within the last 12 months
2. Cardiac status New York Heart Association (NYHA) III-IV
3. Impaired renal function as shown by, but not limited to, serum creatinine ≥ 1.5 mg/dL for males, or ≥ 1.4 mg/dL for females
4. Chronic use of insulin: (more than 3 weeks of continuous use) in the past 12 months
5. Acute infection
6. Clinically significant peripheral edema
7. Acute or chronic history of metabolic acidosis, including diabetic ketoacidosis
8. Clinical evidence of active liver disease, or serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 2.5 times the upper limit of the normal range
9. History of hypoglycemia unawareness
10. Pregnancy or lactation
11. Known hypersensitivity to insulin glargine or any of the components of Lantus®
12. Known hypersensitivity to insulin glulisine or any of the components of Apidra®
13. Any malignancy within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or adequately treated cervical carcinoma in situ
14. Current addiction or current alcohol abuse, or history of substance or alcohol abuse within the last 2 years
15. Diagnosis of dementia
16. Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
17. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study. Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
18. subject is currently taking or was treated with the following medications 3 months prior to screening: Byetta(exenatide), Starlix(nateglinide),Prandin (repaglinide), Januvia(sitagliptin), Janumet(metformin + sitagliptin)
19. Any disease or condition that in the opinion of the investigator and/or sponsor may interfere with the completion of the study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2006-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Jean-Louis, Study Director — Sanofi
Locations (1):
- sanofi-aventis, US, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD): Arm 1: Insulin glargine (IG) administered subcutaneously once daily plus a sulfonylurea and a TZD. Insulin glulisine will be added after Week 12 or later for those subjects needing prandial insulin therapy (HbA1c >6.5%)
- Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD): Arm 2: Insulin glargine (IG) administered subcutaneously once daily plus metformin and a TZD. Insulin glulisine will be added after Week 12 or later for those subjects needing prandial insulin therapy (HbA1c >6.5%)
- Insulin Glargine + Metformin (MET) + Sulfonylurea (SU): Arm 3: Insulin glargine (IG) administered subcutaneously once daily plus metformin and a sulfonylurea. Insulin glulisine will be added after Week 12 or later for those subjects needing prandial insulin therapy (HbA1c >6.5%)
Period: Overall Study
Arm/Group | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU)
Started | 128 (2 randomized patients did not receive study drug and were not included in the safety population) | 128 (1 randomized patient did not receive study drug and was not included in the safety population) | 130 (1 randomized patient did not receive study drug and was not included in the safety population)
Completed | 70 | 83 | 76
Not Completed | 58 | 45 | 54
Not completed — Adverse Event | 6 | 1 | 4
Not completed — Protocol Violation | 3 | 0 | 3
Not completed — Death | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Lost to Follow-up | 4 | 2 | 5
Not completed — Withdrawal by Subject | 26 | 24 | 19
Not completed — Discontinuation of Study | 18 | 16 | 20
Not completed — No longer requires study treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SU + TZD + IG: Arm 1: Insulin glargine(IG) administered subcutaneously once daily plus a sulfonylurea and a thiazolidinedione(TZD). Insulin glulisine will be added after Week 12 or later for those subjects needing additional prandial insulin therapy (HbA1c >6.5%)
- MET + TZD + IG: Arm 2: Insulin glargine (IG) administered subcutaneously once daily plus metformin and a thiazolidinedione (TZD). Insulin glulisine will be added after Week 12 or later for those subjects needing additional prandial insulin therapy (HbA1c >6.5%)
- MET+SU + IG: Arm 3: Insulin glargine (IG) administered subcutaneously once daily plus metformin and a sulfonylurea. Insulin glulisine will be added after Week 12 or later for those subjects needing additional prandial insulin therapy (HbA1c >6.5%)
- Total: Total of all reporting groups
Arm/Group | SU + TZD + IG | MET + TZD + IG | MET+SU + IG | Total
Number analyzed (Participants) | 128 | 128 | 130 | 386
Age Continuous [Mean (Standard Deviation); unit: years] | 56.1 (9.57) | 54.7 (10.14) | 54.6 (9.41) | 55.2 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 54 | 52 | 157
  Male | 77 | 74 | 78 | 229
Region of Enrollment [Number; unit: participants]
  USA | 128 | 128 | 130 | 386
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 33.2 (6.41) | 34.3 (6.57) | 34.5 (7.04) | 34.0 (6.69)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 10.5 (6.95) | 9.7 (5.68) | 10.5 (6.00) | 10.2 (6.23)
Weight [Mean (Standard Deviation); unit: kg] | 98.1 (21.46) | 99.6 (20.22) | 101.2 (24.98) | 99.6 (22.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c) From Baseline to Week 12
Time Frame: 12 weeks from Baseline
Population: Safety Population (excluding patients from Good Clinical Practice [GCP] non-compliant sites)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU)
Number analyzed (Participants) | 116 | 111 | 120
Percentage | -1.2 (1.72) | -1.2 (1.35) | -1.2 (1.31)

2. Secondary Outcome: Change From Baseline to Individual Time Points in HbA1c, Insulin Doses, and Total Insulin Dosage
Time Frame: 60 weeks from Baseline
Population: The study was terminated prematurely due to technical issues with electronic diary data. Consequently, some of the initially planned efficacy analyses, based directly or indirectly on the e-diary data, were not performed.
Measure: Number; unit: Percentage
Arm/Group | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Subjects Achieving an HbA1C Less Than (<) 7.0% and Less Than (<) 6.5%
Time Frame: 60 weeks from Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline to Study Time Points in 7-point Blood Glucose (BG) Profile (Before Meals, 2 Hours After Meals, at Bedtime)
Time Frame: 60 weeks from Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU)
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline to End of Study and to Individual Time Points in Components of Lipid Profile (Total Cholesterol, High-density Lipoprotein Cholesterol [HDL], Low-density Lipoprotein Cholesterol [LDL], Triglycerides, LDL Subfractions)
Time Frame: 60 weeks from Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Occurrences of Hypoglycemia, Symptomatic Hypoglycemia, Severe Hypoglycemia, and Serious Hypoglycemia
Description: * Symptomatic hypoglycemia (BG<70 mg/dL, BG<50 mg/dL): including 1 or more symptoms: headache, dizziness, general feeling of weakness, drowsiness, confusion, pallor, irritability, trembling, sweating, rapid heartbeat & a cold, clammy feeling.
  * Mild-to-moderate hypoglycemia: SMBG ≥ 36 mg/dL but <70 mg/dL
  * Severe hypoglycemia: assistance of another party is required & either:
    * SMBG of <36 mg/dL, or
    * with prompt response to treatment with oral carbohydrates, IV glucose or glucagon.
  * Serious hypoglycemia:
    * Hypoglycemia with coma/loss of consciousness Or Hypoglycemia seizure/convulsion.
Time Frame: 60 weeks from Baseline
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU)
Number analyzed (Participants) | 128 | 128 | 130
Participants
  Any reported symptomatic Hypoglycemic event | 110 | 107 | 112
  Symptomatic events with Self-monitored BG (SMBG) | 109 | 106 | 112
  SMBG <70 mg/dL with symptom | 107 | 102 | 112
  SMBG <50mg/dL with symptom | 74 | 71 | 85
  SMBG <36 mg/dL with symptom | 23 | 24 | 35
  Severe Hypoglycemias | 8 | 10 | 5
  Severe only due to SMBG <36mg/dL | 1 | 1 | 0
  Severe: Prompt response to CHO countermeasure | 4 | 5 | 4
  Severe:SMBG<36mg/dL, prompt response to CHO | 3 | 4 | 2
  Serious hypoglycemia | 3 | 1 | 0
  Coma/Loss of Consciousness | 3 | 1 | 0

7. Secondary Outcome: Rate of Hypoglycemia, Symptomatic Hypoglycemia, Severe Hypoglycemia and Serious Hypoglycemia
Description: as for outcome 6
Time Frame: 60 Weeks from Baseline
Population: Safety Population
Measure: Mean (Standard Deviation); unit: events/ patient-year
Arm/Group | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU)
Number analyzed (Participants) | 128 | 128 | 130
events/ patient-year
  Exposure (Patient-years) | 0.941 (0.3285) | 0.943 (0.3692) | 0.967 (0.3118)
  Hypoglycemic (HE) event with SMBG <70mg/dL | 30.1 (35.54) | 16.5 (20.35) | 25.3 (26.81)
  HE with SMBG <50mg/dL | 4.9 (7.48) | 3.3 (5.74) | 5.6 (8.17)
  HE with SMBG <36mg/dL | 0.3 (0.87) | 0.3 (0.76) | 0.6 (1.55)
  Severe HE (BG<36mg/dL or prompt response to CHO | 0.1 (0.31) | 0.1 (0.53) | 0.1 (0.30)
  Serious HE (coma/loss of consciousness,seizure) | 0.0 (0.14) | 0.0 (0.09) | 0.0 (0.00)

ADVERSE EVENTS:
Arm/Group | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU)
Serious Adverse Events (participants affected / at risk) | 22/128 | 20/128 | 13/130
Other Adverse Events (participants affected / at risk) | 99/128 | 84/128 | 84/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) (N=128) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) (N=128) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU) (N=130)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 3 | 2 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 5 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 2 | 0 | 0
Myelitis transverse (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Arterial stenosis (Vascular disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine + Sulfonylurea (SU) + Thiazolidinedione (TZD) (N=128) | Insulin Glargine + Metformin (MET) + Thiazolidinedione (TZD) (N=128) | Insulin Glargine + Metformin (MET) + Sulfonylurea (SU) (N=130)
Nasopharyngitis (Infections and infestations) | 11 | 12 | 14
Upper respiratory tract infection (Infections and infestations) | 9 | 17 | 9
Bronchitis (Infections and infestations) | 11 | 7 | 6
Influenza (Infections and infestations) | 6 | 7 | 7
Sinusitis (Infections and infestations) | 7 | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 6 | 7 | 5
Weight increased (Investigations) | 8 | 3 | 1
Edema Peripheral (General disorders) | 16 | 6 | 11
Hypertension (Vascular disorders) | 4 | 2 | 7

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to technical issues with electronic diary data. Consequently, some of the initially planned efficacy analyses, based directly or indirectly on the e-diary data, were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.